CLINICAL TRIAL: NCT06845267
Title: Chrono-behavioral Therapy for Chronic Fatigue in Cancer
Acronym: ChronoBT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Lisa Maria Wu, Principal Investigator, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChronoBT
Record Dates: First submitted 2025-02-17; First posted 2025-02-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Chronic Fatigue; Cancer Survivors
MeSH Terms: interventions — Chronotherapy

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned to one of eight 4-week intervention conditions to test the optimal combination of the three ChronoBT components utilizing a Multiphase Optimization Strategy (MOST).
Masking Description: The researcher in charge of the randomization is masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Condition A: light/dark, eating and activity (Experimental): Condition A: light/dark, eating and activity:
  Bright white light glasses 30 minutes upon awakening and blue light blocking glasses 3 hours before bedtime; eating within a 10-hour window, and taking a 15 minutes daily walk.
  Interventions: Behavioral: Chronotherapy
- Condition B: Light/dark and eating (Experimental): Condition B: Light/dark and eating:
  Bright white light glasses 30 minutes upon awakening and blue light blocking glasses 3 hours before bedtime and eating within a 10-hour window.
  Interventions: Behavioral: Chronotherapy
- Condition C: Light/dark and activity (Experimental): Condition C: Light/dark and activity:
  Bright white light glasses 30 minutes upon awakening and blue light blocking glasses 3 hours before bedtime and taking a 15 minutes daily walk.
  Interventions: Behavioral: Chronotherapy
- Condition D: Eating and activity (Experimental): Condition D: Eating and activity:
  Eating within a 10-hour window and taking a 15 minutes daily walk.
  Interventions: Behavioral: Chronotherapy
- Condition E: Light/dark (Experimental): Condition E: Light/dark:
  Bright white light glasses 30 minutes upon awakening and blue light blocking glasses 3 hours before bedtime
  Interventions: Behavioral: Chronotherapy
- Condition F: Eating (Experimental): Condition F: Eating:
  Eating within a 10-hour window
  Interventions: Behavioral: Chronotherapy
- Condition G: Activity (Experimental): Condition G: Activity:
  Taking a15 minutes daily walk.
  Interventions: Behavioral: Chronotherapy
- Condition H: Circadian watch (Active Comparator): Condition H: Circadian watch:
  Waring a circadian watch to access circadian activity
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Chronotherapy — This study utilize and test different combinations of three types of interventions (zeitgebers) to entrain the circadian rhythm: 1) Light being the primary photic zeitgebers that directly entrain the SCN, 2) physical activity and 3) timing of eating) being non-photic zeitgebers that drive peripheral rhythms.
  Arms: Condition A: light/dark, eating and activity; Condition B: Light/dark and eating; Condition C: Light/dark and activity; Condition D: Eating and activity; Condition E: Light/dark; Condition F: Eating; Condition G: Activity
Behavioral: Control — Control condition
  Arms: Condition H: Circadian watch

SUMMARY:
Cancer-related fatigue (CRF) is a severe and persistent side effect of cancer and its treatment, affecting up to 40% of patients and significantly reducing quality of life. Recent research suggests that circadian rhythm disruption has been implicated as a possible related pathophysiological mechanism underlying CRF. Circadian rhythms are 24-hour cycles regulating physiology and behavior through environmental cues called "zeitgebers." Strengthening these cues-such as light exposure, physical activity, and eating-may help reduce CRF.

This project will develop and test the optimal combination a home-based, low-burden chrono-behavioral therapy (ChronoBT) targeting these zeitgebers.

DETAILED DESCRIPTION:
Cancer-related fatigue (CRF) is frequently reported as the most severe and distressing side effect of cancer and its treatment. Among cancer patients, up to 40% will experience CRF that can last months or even years after treatment and it is also deleterious to quality of life. However, there is still no established CRF treatment. Underlying mechanisms of CRF are likely multi-factorial and recently, circadian rhythm disruption has been implicated as a possible related pathophysiological mechanism underlying CRF. Circadian rhythms are endogenous 24-hour cycles of rhythmicity in physiology and behavior orchestrated by the suprachiasmatic nuclei (SCN) in the brain. They are entrained to the environment via time-giving cues called "zeitgebers". Thus, improving circadian rhythm robustness by strengthening modifiable zeitgebers is one potential way to ameliorate CRF. The overarching goal of the proposed project is to conduct an optimization trial of a home-based, low-burden multicomponent chrono-behavioral therapy (ChronoBT) that aims to strengthen the effects of 3 zeitgebers to treat CRF - light/dark exposure, physical activity and eating - all of which individually have shown promise in strengthening circadian rhythms and reducing fatigue. The study will include two work packages: In Work Package 1 (WP1), the investigators will pilot test candidate intervention components in prostate and female breast cancer survivors. In Work Package 2 (WP2), a fully powered optimization trial will be undertaken using the framework - the Multiphase Optimization Strategy (MOST), to test the optimal combination of ChronoBT components.

ELIGIBILITY:
Inclusion Criteria:

1. prostate or female breast cancer survivors
2. completed local and/or adjuvant cancer therapy (with the exception of hormonal therapy) ≥ 1 year previously
3. ≥18 years of age
4. able to speak and read Danish
5. experiencing CRF (score ≤36 on FACT-F)

Exclusion Criteria:

1. use of light therapy in the last year
2. confounding underlying medical/psychiatric disorders or use of medications associated with fatigue (e.g., a central nervous system cancer, untreated hypothyroidism, anemia, chronic fatigue syndrome, insomnia, major depression)
3. non-cancer related factor likely to be a driver of fatigue (e.g., shift work, pregnancy, recent travel across time zones)
4. recurrence of cancer or new cancer
5. physical or psychological conditions that could prevent participation in intervention components
6. use of photosensitizing medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Cancer-related Fatigue | T1 (Baseline, pre-intervention), T2 (two weeks post intervention initiation), T3 (1 day post intervention completion), T4 (follow-up 4 weeks post intervention completion)
  Cancer-related Fatigue by the Functional Assessment of Cancer Therapy - Fatigue Scale (FACT-F) Number of items: 13. Score range: 0-52. Lower score indicates more fatigue.

SECONDARY OUTCOMES:
Sleep Quality | T1 (Baseline, pre-intervention), T2 (two weeks post intervention initiation), T3 (1 day post intervention completion), T4 (follow-up 4 weeks post intervention completion)
  Sleep quality by the Pittsburg Sleep Quality Index (PSQI), measuring seven domains. Higher score indicates worse sleep.
Insomnia | T1 (Baseline, pre-intervention), T2 (two weeks post intervention initiation), T3 (1 day post intervention completion), T4 (follow-up 4 weeks post intervention completion)
  Insomnia by the Insomnia Severity Index (ISI). Number of items: 7. Score range: 0-28. Higher score indicate worse insomnia.
Anxiety and Depression | T1 (Baseline, pre-intervention), T2 (two weeks post intervention initiation), T3 (1 day post intervention completion), T4 (follow-up 4 weeks post intervention completion)
  Anxiety and Depression by the Hospital Anxiety and Depression Scale (HADS). Number of items: 14. Score range: 0-21 for each domain. Higher score indicates worse symptoms.
Health-related Quality of Life | T1 (Baseline, pre-intervention), T2 (two weeks post intervention initiation), T3 (1 day post intervention completion), T4 (follow-up 4 weeks post intervention completion)
  Health-related Quality of Life by the Functional Assessment of Cancer Therapy - General (FACT-G). Number of items: 27. Score range: 0-128. Higher score indicates worse quality of life.
Cognition | T1 (Baseline, pre-intervention), T2 (two weeks post intervention initiation), T3 (1 day post intervention completion), T4 (follow-up 4 weeks post intervention completion)
  Quality of Life - Cognition items from the European Organization for Research and Treatment of Cancer Questionnaires (EORTC-QLQ-30). Number of items: 2. Score range: 2-8. Higher score indicate more impairment.
Circadian Function | During the entire period of intervention and follow-up T4 (4 weeks post intervention completion)
  Circadian Function Index derived from actigraphy data. Score range: 0-1. Higher score indicate more robust rhythms.
Chronotype | T1 (Baseline)
  Chronotype by the reduced Morningness-Eveningness Questionnaire (rMEQ). Number of items: 5. Score range 5-25. Higher score indicates closer to morningness type, while lower score indicate closer to eveningness type.
Credibility/Expectancy | T1 (Baseline)
  Credibility/Expectancy by the Credibility/Expectancy Questionnaire (CEQ). Number of items: 6. Item score range: 1-9. Higher score indicates more credibility/expectancy.
Treatment Satisfaction | T3 (1 day post intervention completion), T4 (follow-up 4 weeks post intervention completion)
  Treatment Satisfaction by the Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General (FACIT-TS-G).
  Number of items: 8. Score range: 0-21. Higher score indicates better satisfaction.

OTHER OUTCOMES:
Adherence and fidelity | During the intervention period: One week for WP1, and four weeks for WP2
  Start/end times of component(s) and protocol deviations by personal logs

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Wu, PhD, Principal Investigator — University of Aarhus; Ali Amidi, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University and Aarhus University Hospital, Aarhus, Denmark